CLINICAL TRIAL: NCT05470660
Title: The Effect of Coronally Advanced Flap With Acellular Dermal Matrix (Alloderm) Versus Coronally Advanced Flap With Micro-needling on RT1 Gingival Recession: A Pilot Study
Brief Title: Coronally Advanced Flap With Alloderm Versus Coronally Advanced Flap With Micro-needling on RT1 Gingival Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Ossama Ezzat Moursy, principle investigator. Salma Ezzat, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER331
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Gingival Recession; Recession, Gingival; Thin-gingiva
Keywords: RT1; Recession; micro-needling; micro-needles; Coronally Advanced Flap; Alloderm
MeSH Terms: conditions — Gingival Recession | interventions — Alloderm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root coverage using coronally advanced flap combined with micro-needling (Experimental): modified coronally advanced flap will be performed in sites of recession defects, then micro-needling will be performed after 1 month from the coronally advanced flap procedure to ensure the initial flap healing
  Interventions: Procedure: Root coverage using coronally advanced flap combined with micro-needling
- coronally advanced flap combined with Alloderm (Active Comparator): modified coronally advanced flap will be performed in sites of recession defects in Association with alloderm to cover the exposed root and 3 mm of connective tissue mesial and distal to it.
  Interventions: Procedure: coronally advanced flap combined with Alloderm

INTERVENTIONS:
Procedure: Root coverage using coronally advanced flap combined with micro-needling — modified coronally advanced flap will be performed in sites of recession defects, then micro-needling will be performed after 1 month from the coronally advanced flap procedure to ensure the initial flap healing.
  Arms: Root coverage using coronally advanced flap combined with micro-needling
Procedure: coronally advanced flap combined with Alloderm — modified coronally advanced flap will be performed in sites of recession defects in Association with alloderm to cover the exposed root and 3 mm of connective tissue mesial and distal to it.
  Arms: coronally advanced flap combined with Alloderm

SUMMARY:
This study aims to assess the effect of micro-needling together with coronally advanced flap procedure on the gain of gingival thickness (GT) and keratinized tissue width (KTW) and compare it to Alloderm with coronally advanced flap procedure in the management of thin periodontal phenotype associated with recession type 1 (RT1)

DETAILED DESCRIPTION:
Gingival or periodontal diseases were found to occur more likely in patients with a thin gingival biotype. The periodontal phenotype was also found to show stronger correlation with gingival thickness rather than keratinized tissue width and papilla height. Moreover, the thin gingiva was usually found to be associated with thin bony plate with potential for dehiscence and fenestration and hence was thought to be at risk for recession after trauma.

Several techniques have been recommended for the treatment of gingival recession. One of the most predictable outcome is associated with the use of a coronally advanced flap and acellular dermal matrix graft.

Treatment of thin periodontal phenotype through the conjunction of i-PRF and micro-needling may be a first move of the non-surgical approach for improving the gingival thickness. Micro-needling was proved to be generally an effective and safe therapeutic option for numerous dermatologic conditions as clinical improvement of scars, striae, and rhytids with appropriate recovery and limited side effects. The controlled dermal wounding and stimulation of the wound healing cascade through Micro-needling was found to enhance collagen production and thus was responsible for the clinical results obtained.

Therefore, this study will be aiming to compare the effect of micro-needling on the gingival thickness in root coverage procedures. It will also provide an insight of its effect on the patient related factors and the root coverage parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patient consulting in the outpatient clinic.

  * Able to tolerate the study procedures.
  * Patient ready to perform oral hygiene instructions.
  * Compliance with the maintenance program.
  * Provide informed consent.
  * Accepts the 6 months follow-up period
* Mature permanent tooth.
* Full-mouth plaque index (PI) and full-mouth bleeding on probing (BOP) score of ≤ 15%.
* Presence of identifiable Cemento-enamel Junction.
* RT1 facial recession defect of ≥3 mm.
* Clinical indication and/or patient request for recession coverage

Exclusion Criteria:

* Medically compromised patients.

  * use of any drugs that might lead to gingival enlargement
  * Pregnant or nursing women.
  * Uncooperative patients.
  * Smokers.
* Teeth with malocclusion, crowding, fillings, missing or supernumerary mandibular anterior teeth.

  * Cairo Recession Type 3 (RT3) recession defects.
  * Teeth with active orthodontic treatment.
  * Previous periodontal surgery.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Gingival thickness (GT) in mm | 6 months
  Gingival thickness (GT) will be specified at a mid-buccal location approximately 1 mm apical to the probing depth (PD) level with a #15 endodontic spreader. The reamer will be pierced, perpendicularly to the mucosal surface, through the soft tissue with light pressure until a hard surface is felt. The silicone disk stop will then be placed in tight contact with the soft tissue surface and fixed by a drop of cyanoacrylate adhesive; after careful removal of the reamer, penetration depth will be measured with a caliper to the nearest 0.1 mm gingival thickness changes will be calculated after 6 months

SECONDARY OUTCOMES:
Keratinized tissue width (KTW) in mm | 6 months
  Keratinized tissue (KT) will be measured from the most apical point of the gingival margin to the mucogingival junction measurements will be recorded at baseline and after 6 months
Clinical Attachment Level (CAL) in mm | 6 months
  Will be measured from the Cemento-enamel Junction to the bottom of the gingival sulcus at baseline and 6 months
Gingival Recession Depth (RD) in mm | 6 months
  Will be measured from the Cemento-enamel Junction to the most apical extension of the gingival margin.
Gingival Recession Width (RW) in mm | 6 months
  Will be measured horizontally between the borders of the recession at the level of Cemento-enamel Junction.
Percentage of root coverage | 6 months
  Preoperative vertical recession - Postoperative vertical recession/preoperative vertical recession) x 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alster TS, Graham PM. Microneedling: A Review and Practical Guide. Dermatol Surg. 2018 Mar;44(3):397-404. doi: 10.1097/DSS.0000000000001248. PMID 28796657
- [Background] Cairo F, Pagliaro U, Nieri M. Treatment of gingival recession with coronally advanced flap procedures: a systematic review. J Clin Periodontol. 2008 Sep;35(8 Suppl):136-62. doi: 10.1111/j.1600-051X.2008.01267.x. PMID 18724847
- [Background] Cortes Ade Q, Martins AG, Nociti FH Jr, Sallum AW, Casati MZ, Sallum EA. Coronally positioned flap with or without acellular dermal matrix graft in the treatment of Class I gingival recessions: a randomized controlled clinical study. J Periodontol. 2004 Aug;75(8):1137-44. doi: 10.1902/jop.2004.75.8.1137. PMID 15455743